CLINICAL TRIAL: NCT06852651
Title: The Efficacy of Superficial Cervical Block Application in Postoperative Analgesia Management in Patients Undergoing Total Laryngectomy and Bilateral Neck Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Hilal AKCA, M.D., Başakşehir Çam & Sakura City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Superficial Cervical Block
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Laryngeal Neoplasm
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Postoperative pain assessments (NRS scores at 30 min, 4 h, 8 h, and 24 h), opioid consumption, and recovery outcomes will be recorded by an independent investigator who is unaware of the intervention status to reduce observer bias.
  Data Analyst Masking:
  The data will be analyzed by a statistician who is blinded to the group assignments to prevent bias in statistical interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial Cervical Block (SCB) Group (Experimental): Patients undergoing total laryngectomy and bilateral neck dissection who receive a superficial cervical block (SCB) for postoperative pain management.
  The block will be performed bilaterally under ultrasound guidance using 0.1 mL/kg of 0.25% bupivacaine after anesthesia induction.
  Postoperative pain scores, opioid consumption, ventilation status, ICU and hospital length of stay, and complications will be recorded.
  Interventions: Procedure: Superficial Cervical Block (SCB) Group
- Control Group (No Block) (No Intervention): Patients undergoing total laryngectomy and bilateral neck dissection who receive standard postoperative analgesia without a superficial cervical block (SCB).
  Postoperative pain management will consist of intravenous analgesics as per institutional protocols.
  The same postoperative parameters (pain scores, opioid use, ventilation status, ICU/hospital stay, and complications) will be assessed for comparison.

INTERVENTIONS:
Procedure: Superficial Cervical Block (SCB) Group — Patients in this group will receive a bilateral superficial cervical block under ultrasound guidance after anesthesia induction but before the surgical procedure begins.
  The block will be performed using 0.1 mL/kg of 0.25% bupivacaine per side, targeting the superficial branches of the cervical plexus.
  The primary goal is to assess its efficacy in postoperative pain management and its impact on recovery parameters.
  Arms: Superficial Cervical Block (SCB) Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of the superficial cervical block in postoperative pain management for patients undergoing total laryngectomy and bilateral neck dissection. It will also assess its impact on recovery and clinical outcomes. The main questions it aims to answer are:

Does the superficial cervical block reduce postoperative pain scores? What are the effects of the block on ventilation status, ICU stay, and hospital length of stay? Researchers will compare patients who receive the superficial cervical block to those who do not, assessing its effectiveness in pain management and postoperative recovery.

Participants will:

Receive a superficial cervical block or standard pain management during surgery Have their pain levels assessed using the Numeric Rating Scale (NRS) at 30 min, 4, 8, and 24 hours postoperatively Have their postoperative ventilation status, ICU stay, hospital length of stay, and complications recorded

DETAILED DESCRIPTION:
Background and Rationale:

Total laryngectomy with bilateral neck dissection is a major head and neck surgery that significantly impacts postoperative recovery and pain management. Effective analgesia is crucial in these patients to facilitate early rehabilitation, optimize respiratory function, and improve overall outcomes. Conventional postoperative pain management strategies often rely on systemic opioids, which may lead to adverse effects such as respiratory depression, nausea, and sedation, potentially delaying recovery and increasing ICU length of stay.

The superficial cervical block (SCB) is a regional anesthesia technique that provides analgesia by targeting the superficial branches of the cervical plexus. It has been shown to reduce postoperative pain in head and neck surgeries while minimizing opioid-related side effects. However, its efficacy in patients undergoing total laryngectomy with bilateral neck dissection remains understudied. This study aims to evaluate whether the addition of a superficial cervical block to standard anesthesia protocols improves postoperative pain management and enhances recovery outcomes in these patients.

Study Objectives:

The primary objective of this study is to determine the effectiveness of the superficial cervical block in reducing postoperative pain in patients undergoing total laryngectomy and bilateral neck dissection.

The secondary objectives include:

Ventilation outcomes: Assessing whether the use of SCB reduces the need for postoperative ventilatory support, including prolonged mechanical ventilation or re-intubation.

ICU admission and hospital length of stay: Evaluating if SCB contributes to shorter ICU and hospital stays by improving pain control and facilitating early mobilization.

Postoperative recovery metrics: Investigating the impact of SCB on post-extubation respiratory function, tracheostomy adaptation, and overall postoperative morbidity.

Opioid consumption: Comparing opioid requirements in patients who receive SCB versus those who do not.

Complication rates: Monitoring for any adverse effects related to SCB, including local anesthetic toxicity, hematoma, or block failure.

Study Design:

This study is designed as a prospective observational trial conducted at a tertiary care hospital. Patients scheduled for total laryngectomy with bilateral neck dissection will be enrolled after obtaining informed consent.

Patient Selection Criteria:

Inclusion Criteria:

Patients undergoing total laryngectomy and bilateral neck dissection. Aged ≥18 years. ASA classification I-IV. Patients who provide written informed consent.

Exclusion Criteria:

Patients undergoing emergency total laryngectomy. Patients with allergy to local anesthetics. Patients with coagulopathy or contraindications to regional anesthesia.

Intervention and Methodology:

All patients will undergo standardized general anesthesia with ASA monitoring, including:

Electrocardiography (ECG) Non-invasive blood pressure monitoring End-tidal CO₂ (EtCO₂) and SpO₂ monitoring Invasive arterial blood pressure monitoring (if required)

After anesthesia induction and orotracheal intubation, patients will be divided into two groups based on anesthesiologist discretion:

SCB Group: Patients will receive an ultrasound-guided superficial cervical block using 0.1 mL/kg of 0.25% bupivacaine bilaterally.

Control Group: Patients will undergo standard postoperative pain management without regional anesthesia.

Postoperative Pain and Recovery Assessments:

Pain assessment: Postoperative pain scores will be recorded using the Numeric Rating Scale (NRS, 0-10) at 30 minutes, 4 hours, 8 hours, and 24 hours postoperatively.

Cough assessment: Cough severity will be graded on a 0-4 scale at the same time points.

Postoperative ventilation status: Duration of mechanical ventilation and incidence of postoperative respiratory complications will be noted.

ICU and hospital stay duration: The total length of ICU and hospital stay will be compared between groups.

Postoperative opioid consumption: The total amount of rescue analgesics (morphine, tramadol, etc.) will be recorded.

Morbidity and mortality: Postoperative complications, including cardiovascular, pulmonary, and surgical site complications, will be documented.

Outcome Measures:

Primary Outcome:

Postoperative pain scores (NRS) at 30 min, 4 h, 8 h, and 24 h.

Secondary Outcomes:

Duration of postoperative ventilation (mechanical ventilation hours, need for reintubation).

ICU and hospital length of stay (days spent in ICU and hospital). Postoperative opioid consumption (total morphine-equivalent dose). Cough severity scores at multiple time points. Postoperative morbidity and mortality rates.

Statistical Analysis Plan:

Categorical data (e.g., ventilation status, ICU admission, mortality) will be analyzed using Chi-square or Fisher's exact test.

Continuous variables (e.g., pain scores, opioid consumption, hospital stay) will be compared using independent samples t-test or Mann-Whitney U test, depending on normality distribution.

Repeated measures analysis (ANOVA or Friedman test) will be applied to assess changes in pain and cough scores over time.

Significance and Impact of the Study:

This study will provide critical insights into the role of superficial cervical block in improving pain control and recovery outcomes in patients undergoing major head and neck surgery.

If effective, SCB may become a standardized part of perioperative pain management in these patients, reducing opioid dependence and enhancing early postoperative recovery.

Findings from this research will be disseminated through peer-reviewed journals and international conferences to contribute to the growing body of evidence supporting regional anesthesia techniques in head and neck surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total laryngectomy with bilateral neck dissection.
* Age ≥18 years.
* ASA (American Society of Anesthesiologists) classification I-IV.
* Patients who provide written informed consent.

Exclusion Criteria:

* Patients undergoing emergency surgery.
* Patients with known allergies to local anesthetics (e.g., bupivacaine, lidocaine).
* Patients with coagulopathy or bleeding disorders that contraindicate regional anesthesia.
* Patients with severe cognitive impairment affecting informed consent.
* Patients with infection at the injection site preventing SCB administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores (NRS) | 30 minutes, 4 hours, 8 hours, and 24 hours postoperatively
  Pain will be assessed using the Numeric Rating Scale (NRS, 0-10) at predefined time points.

SECONDARY OUTCOMES:
Postoperative Opioid Consumption | 1 day
  Total morphine-equivalent opioid usage will be recorded.
Cough Severity Score | 30 minutes, 4 hours, 8 hours, and 24 hours postoperatively
  Cough severity will be graded on a 0-4 scale (0 = no cough, 4 = severe cough affecting recovery).

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir cam and sakura city hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided